CLINICAL TRIAL: NCT06310629
Title: Comparison of Oxygenation Efficacy of "Intrinseque Health" Non-Rebreathing Mask ("IHNRM") vs. High Flow Nasal Cannula (HFNC)
Brief Title: Oxygenation Efficacy of "Intrinseque Health" Non-Rebreathing Mask ("IHNRM")
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMUH112-REC3-163
Record Dates: First submitted 2024-02-21; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Disease; Respiratory Distress Syndrome; Respiratory Failure
Keywords: SpO2、extubation、EtCO2
MeSH Terms: conditions — Respiration Disorders; Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Flow Nasal Cannula (Active Comparator): High Flow Nasal Cannula
  Interventions: Device: High Flow Nasal Cannula
- "Intrinseque Health" Non-Rebreathing Mask ("IHNRM") (Experimental): "Intrinseque Health" Non-Rebreathing Mask ("IHNRM")
  Interventions: Device: "Intrinseque Health" Non-Rebreathing Mask ("IHNRM")

INTERVENTIONS:
Device: High Flow Nasal Cannula — High Flow Nasal Cannula
  Arms: High Flow Nasal Cannula
Device: "Intrinseque Health" Non-Rebreathing Mask ("IHNRM") — "Intrinseque Health" Non-Rebreathing Mask ("IHNRM")
  Arms: "Intrinseque Health" Non-Rebreathing Mask ("IHNRM")

SUMMARY:
Based on early bench-testing data and subsequent clinical case studies in the U.S., "Intrinseque Health" non-rebreathing mask (IHNRM) has delivered virtual elimination of air entrainment and preferential delivery of all available oxygen first into the alveolar spaces by sequential opening of valves in its controller manifold, even at oxygen flow as low as 10 LPM, patient can attain high alveolar oxygen concentration of 75% or more-far higher than attainable with face mask or nasal cannula.

Numerous intubated patients emerging from the operating room require intensive critical care specialist supervision in order to transition to the regular care. This would enable higher patient turnover and more efficient utilization of hospital resources, if patient can be transited to the regular care earlier by using a device that supports high oxygenation. This will enable a faster, safe and smooth extubation in critical care, and earlier discharge from intensive care ward.

This study is anticipated to take only around 2.5 hour per patient to complete. Patients meeting the inclusion and exclusion criteria of this study are placed on IHNRM and monitored until steady state of SpO2 of 95% or higher on 7-10 LPM has been maintained for at least 2 hours, when they can be discharged from the post-anesthesia care unit (PACU) to the regular care ward.

The study is the parallel design study. 60 patients will be randomly selected to use the IHNRM, and 30 subjects will be placed on HFNC. Blood oxygen concentration (SpO2), respiratory rate, end tidal CO2 concentration (EtCO2), and vital sign will be recorded in the study. The endpoint of the study is to compare the effect after using between "IHNRM" and HFNC.

ELIGIBILITY:
Inclusion Criteria:

1. ANY hospitalized patient in moderate to moderately severe respiratory distress and able to breathe spontaneously, and with SpO2 (oxygen saturation by pulse oximetry) reading of:

   (i) 90% or less on room air, or (ii) <95% in spite of oxygen supplementation on another form of oxygen supplementation.
2. Has minimum ideal body wt. of at least ≥15 kg., and at least 3 years old.
3. Self/guardian-able to consent to study participation and monitoring.

Exclusion Criteria:

Patient with any of the following present will be excluded:

1. Agitated or confused or somnolent mental state.
2. Any impairment of gag reflex.
3. Multi-organ failure that may decompensate rapidly, with or without hypoperfusion secondary to cardiogenic, hypovolemic, or septic shock.
4. Acute MI, pulmonary embolism, pneumothorax or stroke
5. Inability to pull mask off (or to side of) face in emergency.
6. ICP (intracranial pressure) > 15mmhg. If ICP unknown but clinically may have elevated ICP (such as head trauma or CNS tumor), patient should be excluded.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-05-21 (Estimated)

PRIMARY OUTCOMES:
Time to reach SpO2 Criteria in Run-in | SpO2 will be recorded in every 5 minutes in Run-in phase up to 30 minutes
  Time to attaining SpO2 is by 4 percentage points or more above the baseline SpO2 while on room air or ≥95% .
The percentage of subjects to reach SpO2 Criteria in maintenance | SpO2 will be recorded in every 30 minutes in maintenance phase up to 2 hours
  Comparing % of patients able to maintain target parameters for a continuous duration of 2 hours or more the time of continuous SpO2 reading of 4 points or more above the baseline SpO2 while on room air or SpO2 reading ≥95%

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ching Yen, PhD, Principal Investigator — Professor
Locations (1):
- Department of Internal Medicine, China Medical Univdersity Hospital, Taichung, Taiwan